CLINICAL TRIAL: NCT04094974
Title: The Usefulness of the Combination of Preoperative Assessment of Optic Nerve Sheath Diameter and Heart Rate Variability to Predict Intraoperative Brain Condition in Patients With Supratentorial Tumors
Brief Title: Heartrate Variability and Intraoperative Brain Conditions in Supratentorial Tumors
Status: Completed | Type: Observational
Sponsor: DyAnsys, Inc. (Industry)
Responsible Party: Sponsor
Other Study IDs: CS009
Record Dates: First submitted 2019-09-13; First posted 2019-09-19 (Actual); Last update posted 2021-01-25 (Actual); Status verified 2021-01

CONDITIONS: Supratentorial Brain Tumors
Keywords: Heart rate variability,; supratentorial brain tumors; optic nerve sheath diameter

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Device: ANSiscope — Heart rate variability will be assessed using ansiscope before surgery

SUMMARY:
This study aims to determine the relationship between heart rate variability and intraoperative brain relaxation conditions in patients with brain tumors.

DETAILED DESCRIPTION:
Patients undergoing brain surgery for treatment of brain tumors will be studied to determine the relationship between heart rate variability and intraoperative brain relaxation conditions.

ELIGIBILITY:
Inclusion Criteria:

* Patient aged 18 to 75 years
* ASA(American Society of Anesthesiologists ) I - III
* Patients undergoing surgery for supratentorial tumors
* Glasgow coma scale > 10

Exclusion Criteria:

* Patient aged below 18 and above 75 years.
* Pregnancy
* ASA(American Society of Anesthesiologists) IV-V
* Previous cranial surgery
* Morbid obesity ( BMI>40)
* Ocular injury/ Glaucoma
* Head injury
* Patient on beta blockers, ACE(angiotensin-converting-enzyme) inhibitors, Clonidine
* Diabetes mellitus for more than 5 years

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adult patients of either sex with supratentorial brain lesions who are posted for neurosurgery will be taken as study population. Patients who meet the inclusion criteria and give consent for the study will be included in the study
Sampling Method: Probability Sample
Enrollment: 58 (Actual)
Dates: Start 2019-10-12 (Actual); Primary Completion 2020-10-03 (Actual); Study Completion 2020-10-03 (Actual)

PRIMARY OUTCOMES:
Brain relaxation | 2hours
  1. Tight Brain-the brain surface is jutting out or expanding beyond the craniotomy margins, brain pulsations are not clearly defined.
  2. Brain surface at level of craniotomy margins, Brain pulsations faintly observed
  3. Brain surface just below the surface of craniotomy margin. Brain pulsations well seen.
  4. Brain surface well below the surface of craniotomy margin, well retracted in to the cranial cavity with good brain pulsations.Brain relaxation score will me measured only once. There is no follow up

SECONDARY OUTCOMES:
Hemodynamic Measurement-Heartrate | 2hours
  The change in hemodynamic variable heart rate in beats per minute will be measured through the study period
Hemodynamic Measurement-Bloodpressure | 2hours
  The change in hemodynamic variable blood pressure in mmHg will be measured through the study period

CONTACTS AND LOCATIONS:
Overall Officials: Dr. Mathangi Krishnakumar, MBBS,MD,DM, Principal Investigator — NIMHANS,Bengaluru
Locations (1):
- National Institute of Mental Health and Neurosciences, Bengaluru, Karnataka, India

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Li J, Gelb AW, Flexman AM, Ji F, Meng L. Definition, evaluation, and management of brain relaxation during craniotomy. Br J Anaesth. 2016 Jun;116(6):759-69. doi: 10.1093/bja/aew096. Epub 2016 Apr 27. PMID 27121854
- [Background] Rasmussen M, Bundgaard H, Cold GE. Craniotomy for supratentorial brain tumors: risk factors for brain swelling after opening the dura mater. J Neurosurg. 2004 Oct;101(4):621-6. doi: 10.3171/jns.2004.101.4.0621. PMID 15481716
- [Background] Robba C, Santori G, Czosnyka M, Corradi F, Bragazzi N, Padayachy L, Taccone FS, Citerio G. Optic nerve sheath diameter measured sonographically as non-invasive estimator of intracranial pressure: a systematic review and meta-analysis. Intensive Care Med. 2018 Aug;44(8):1284-1294. doi: 10.1007/s00134-018-5305-7. Epub 2018 Jul 17. PMID 30019201
- [Background] Schmidt EA, Despas F, Pavy-Le Traon A, Czosnyka Z, Pickard JD, Rahmouni K, Pathak A, Senard JM. Intracranial Pressure Is a Determinant of Sympathetic Activity. Front Physiol. 2018 Feb 8;9:11. doi: 10.3389/fphys.2018.00011. eCollection 2018. PMID 29472865
- [Background] Furgala A, Madroszkiewicz D, Madroszkiewicz E, Goscinski I, Kolasinska-Kloch W, Moskala M, Thor PJ. Autonomic system disturbances in patients with increased intracranial pressure caused by brain tumors evaluated by heart rate variability. Folia Med Cracov. 2007;48(1-4):35-44. PMID 19051691
- [Background] Jadhav T, Sriganesh K, Thirthalli J, Reddy KRM, Venkataramaiah S, Philip M, Naveen Kumar C, Armugham SS. Effect of Atropine Premedication on Cardiac Autonomic Function During Electroconvulsive Therapy: A Randomized Crossover Study. J ECT. 2017 Sep;33(3):176-180. doi: 10.1097/YCT.0000000000000417. PMID 28471773
- [Background] Weickenmeier J, Saze P, Butler CAM, Young PG, Goriely A, Kuhl E. Bulging brains. J Elast. 2017 Dec;129(1-2):197-212. doi: 10.1007/s10659-016-9606-1. Epub 2016 Oct 24. PMID 29151668
- [Background] Hernandez-Palazon J, Fuentes-Garcia D, Domenech-Asensi P, Piqueras-Perez C, Falcon-Arana L, Burguillos-Lopez S. A comparison of equivolume, equiosmolar solutions of hypertonic saline and mannitol for brain relaxation during elective supratentorial craniotomy. Br J Neurosurg. 2016;30(1):70-5. doi: 10.3109/02688697.2015.1109061. Epub 2015 Nov 16. PMID 26571037
- [Background] Cold GE, Tange M, Jensen TM, Ottesen S. "Subdural' pressure measurement during craniotomy. Correlation with tactile estimation of dural tension and brain herniation after opening of dura. Br J Neurosurg. 1996 Feb;10(1):69-75. doi: 10.1080/02688699650040548. PMID 8672261